CLINICAL TRIAL: NCT06792799
Title: An Exploratory Clinical Study on the Safety and Efficacy of CD19/BCMA Chimeric Antigen Receptor NK Cells in the Treatment of B Cell-related Autoimmune Diseases in Children
Brief Title: Anti-CD19/BCMA CAR-NK Cells in Patients With B Cell Mediated Autoimmune Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SC-0002-P-01
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases; Systemic Lupus Erthematosus; Multi-Drug Resistant Nephrotic Syndrome; IgAN - IgA Nephropathy
Keywords: car-nk; Multi-Drug Resistant Nephrotic Syndrome; Systemic Lupus Erthematosus; IgAN - IgA Nephropathy
MeSH Terms: conditions — Autoimmune Diseases; Nephrotic Syndrome; Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/BCMA CAR NK cells (Experimental): The study adopted a dose-escalation and expansion study design. All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by anti-CD19/BCMA CAR NK cells infusion.
  Interventions: Biological: anti-CD19/BCMA CAR NK cells (KN5601)

INTERVENTIONS:
Biological: anti-CD19/BCMA CAR NK cells (KN5601) — Patients will receive Fludarabine (30 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3. Multiple doses of anti-CD19/BCMA CAR NK cells (KN5601) will infused in each group using dose-escalation strategy.

SUMMARY:
this is an investigator-initiated trial aimed at evaluating the efficacy and safety of anti-CD19/BCMA CAR-NK Cells in Patients With B cell mediated autoimmune disease.

DETAILED DESCRIPTION:
Autoimmune diseases are conditions in which the immune system fails to accurately recognize normal tissues or cells, leading to the attack of organs, tissues, or cells.

Systemic lupus erythematosus (SLE) is a severe autoimmune disorder that can cause widespread damage to multiple organs and systems, ultimately resulting in disability and even death. Pediatric patients with SLE are particularly susceptible to organ damage, especially renal impairment, and typically experience a more severe and protracted disease course compared to adults. Despite advances in therapy, many patients continue to suffer from SLE. In China, only 0.76% to 25% of patients achieve drug-free or clinical remission, highlighting the urgent need for novel therapeutic approaches.

For patients with multi-drug resistant nephrotic syndrome (MDR-SRNS), who are at high risk of progressing to kidney failure, there remains no effective treatment. Therefore, there is a pressing need for new therapeutic strategies.

Immunoglobulin A nephropathy (IgAN) is the most common primary glomerulonephritis worldwide. Although immunosuppressants have been used in some patients, IgAN remains a leading cause of kidney failure in young adults, with approximately 40% of patients progressing to end-stage kidney disease (ESKD) within 20-30 years.

Since 2019, CAR T-cell therapy has shown success in treating various autoimmune diseases, including SLE, systemic sclerosis, and idiopathic inflammatory dermatomyositis. However, the widespread application of autologous CAR T-cells is limited by several factors, including their high cost and the frequent occurrence of adverse effects. Autologous CAR T-cells are personalized products, which make them expensive and less accessible. Furthermore, the risks of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) remain significant concerns.

Chimeric antigen receptor natural killer (CAR-NK) cell therapy offers a promising alternative. This adoptive cell therapy involves the genetic modification of NK cells to recognize and eliminate target cells expressing disease-related antigens. CAR-NK cells have several advantages over CAR T-cells, including a lower risk of graft-versus-host disease (GVHD) and minimal occurrence of CRS or ICANS. Additionally, CAR-NK therapy is more cost-effective, which could greatly enhance its accessibility.

Given these advantages, CAR-NK cell therapy holds potential for revolutionizing the treatment of refractory SLE and MDR-SRNS, IgAN, offering new hope for patients with these challenging conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians must acknowledge the risks and procedures involved and subsequently provide informed consent to participate in the clinical trial.
2. Predicted survival time ≥ 12 weeks;
3. ECOG: 0~2;
4. Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% ;
5. Renal function: eGFR≥30ML/min/1.73m2； (For patients with an eGFR < 30 mL/min/1.73 m² or those receiving renal replacement therapy, inclusion or exclusion in the study is determined at the discretion of the investigators. )
6. Liver function: Asparagus cochinchinensis transase (AST) and Alanine Aminotransferase (ALT)≤3.0 ULN, Total Bilirubin (TBIL) in serum ≤2.0×ULN;
7. Lung function: No serious lung lesions, SpO2≥92%;
8. Negative pregnancy test for female Subjects of childbearing age, agree to take effective contraceptive measures the first year after CAR-NK infusion;

SLE:

1. Age:≥5 years old;
2. Diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria；
3. Still in moderate to severe disease activity despite ≥3M of high dose glucocorticoids(prednisone≥1mg/kg/d or other equivalent amount of other steriod ), hydroxychloroquine and at least 2 of the following treatments(cyclophosphamide, MMF, azathioprine, methotrexate, cyclosporin, tacrolimus, sirolimus, leflunomide, telitacicept, Beliumab, and rituximab,etc,al); or Intolerant to standard treatments; or the dosage of steroid can not be reduced to 5mg/d after 6-month of routine treatment.
4. SLEDAI 2K score>6 points;
5. No history of Central nervous system (CNS) disease within 60 days prior to screening;
6. No history of macrophage activation syndrome (MAS) within one month prior to screening.

MDR-SRNS

1. Age ≥3 years old, gender unlimited;
2. Diagnosed with SRNS according to the 2021 Kidney Disease: Improving Global Outcomes （KDIGO） Guidelines and have not achieved a complete response after 12 months of treatment with two standard doses of hormone replacement drugs with different mechanisms of action or relapse of disease activity after remission (at least one of the two drugs is a calcineurin inhibitor such as cyclosporine or tacrolimus; Other hormone replacement drugs include Mycophenolate Mofetil, cyclophosphamide, Taitacept or rituximab); Or if no remission has been achieved after 3 to 6 months of adequate treatment with one calcineurin inhibitor, if the researcher judges that the benefits outweigh the risks and the patient or guardian has fully informed consent, the patient can be considered for inclusion.Patients with other diseases, such as systemic lupus erythematosus, requiring long-term systemic treatment with glucocorticoids or immunosuppressants, may be considered for inclusion after the investigator determines that the benefits outweigh the risks and the patient or guardian has fully informed consent;
3. Renal biopsy was performed and the pathological type was determined to be minimal lesion nephropathy(MCD) or focal segmental glomerulosclerosis (FSGS);

IgA nephropathy

1. Age: ≥ 5 years old, male or female;
2. IgA nephropathy pathologically confirmed by renal biopsy;
3. Angiotensin-Converting Enzyme Inhibitors (ACE) or angiotensin receptor blocker (ARB) treated for at least 3 months and meet at least one of the following requirements:

   1. Combination or sequential treatment with steroids and at least one immunosuppressant or biologic for ≥ 3 months; and 24-hour urine protein quantification ≥500mg or UPCR≥0.5mg/mg;
   2. >50% decline in eGFR within 3 months;
   3. Patients who are unable to tolerate conventional treatment and for whom the investigator determines the benefits outweigh the risks and who have obtained fully informed consent from the patient or guardian may be considered for inclusion;
4. Exclude subjects with other secondary causes; exclude patients with uncontrolled blood pressure.

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, obinutuzumab), or subjects with a history of severe allergic reactions
2. Uncontrollable infection, or active infection that requires systemic treatment within 1 week prior to screening；
3. Subjects with grade III or IV heart failure (NYHA classification)
4. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs；
5. Renal replacement therapy has been or is being performed within 3 months prior to transfusion;
6. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
7. Signs of herpes or varicella-zoster virus infection (especially chickenpox, shingles) within 12 weeks prior to screening;
8. Patients had seizure, or other active central nervous system disease;
9. Patients with malignant diseases such as tumors before screening, or with other serious life-threatening diseases;
10. Secondary or congenital immunodeficiency.
11. History of any cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal disease or other major medical condition that would prevent the administration of KN5601, except for lupus (determined by the investigator)
12. Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months prior to screening; Acute graft-versus-host disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening;
13. Received live vaccine within 4 weeks before screening;
14. Subjects who have received B cell-targeted drug therapy within 1 month before enrollment
15. Tested positive in Blood pregnancy test；
16. Patients who participated in other clinical study within 3 months prior to enrollment;
17. Any abnormal laboratory test results judged by the investigator to be clinically significant and prevent the subject from participating in the study. Laboratory test values that are out of range and not of clinical significance will not be considered as exclusion criteria
18. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR-NK cell therapy in patients with B cell mediated autoimmune disease | 1 months
  Incidence of Dose Limiting Toxicity (DLTs), Incidence and severity of Adverse Events (AEs) and Serious Adverse Event（SAEs）.
The efficiency of CAR-NK cell therapy in patients with B cell mediated autoimmune disease | 3 months
  SLE: The rate of patients achieving SRI-4 response, LLDAS, or DORIS remission MDR-SRNS:Complete response and partial response rate. IgAN:partial or complete response.

SECONDARY OUTCOMES:
Effectiveness of other visit points | 6 months
  The responsive rate and the rate of complete /partial remission

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang 310000, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No